CLINICAL TRIAL: NCT00630136
Title: Effectiveness of the Consent Process Used for Outpatient Endoscopy
Brief Title: Effectiveness of the Consent Process
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Nancy Neilan, MT (ASCP)/ Research Coordinator, Children's Mercy Hospitals and Clinics
Other Study IDs: CMH080104
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2008-10

CONDITIONS: Parental Consent
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Adult parent or legally authorized representative (LAR) of child who has consented to undergo an out-patient endoscopy at Children's Mercy Hospital as a diagnostic procedure
  Interventions: Behavioral: interview

INTERVENTIONS:
Behavioral: interview — The parent/LAR who has consented to have their child undergo an outpatient endoscopy procedure will be interviewed prior to the procedure being performed.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the consent process currently used for outpatient endoscopy procedures at our hospital. Results from this study will be used to assist in making improvements in the way we communicate with parents, thereby enhancing the ability to provide informed consents.

DETAILED DESCRIPTION:
Obtaining informed consent before performing an invasive medical procedure or treatment is a crucial component of patient care. The manner in which the consent process is conducted impacts the doctor/patient relationship, patient safety and patient satisfaction. Many times, patients sign consent forms without reading or understanding them. Although the form has been signed, true informed consent has not been obtained. While there are many variables that impact the ability to truly consent, ineffective communication between the patient and health care providers hampers the process.

Evidence shows that improving the consent process by ensuring effective communication between the child's parent and health care team affords substantial benefit. A consent process well done strengthens the parent-provider relationship. It positively impacts risk management. It improves patient safety. It diffuses would-be litigants by helping parents have realistic expectations of care. The consent process should allow and encourage parents to exercise both their right and their responsibility to take an active role in their child's health care.

ELIGIBILITY:
Inclusion Criteria:

* Adult parent or legally authorized representative (LAR) of child who has consented to undergo an out-patient endoscopy at CMHC as a diagnostic procedure
* Ability to converse in English
* Provided implied consent prior to data collection and verbal consent after data collection to participate in this research study

Exclusion Criteria:

* Any parent/ LAR under the age of 18 years
* Time constraint or verbally stating they do not wish to provide study data prior to child undergoing endoscopy
* Stating they do not wish to have these data used as study data after completion of the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gastroenterology primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
determine if the parent/LAR has an understanding of why the endoscopy procedure has been recommended and what it involves | after obtaining consent for endoscopy but prior to endoscopy procedure
determine if the parent/ LAR has an understanding of the probable benefits and risks associated with endoscopy | after obtaining consent for endoscopy but prior to endoscopy procedure

SECONDARY OUTCOMES:
determine if the parent/LAR knows who will be present during the procedure | after obtaining consent for endoscopy but prior to endoscopy procedure
determine if the parent/LAR has an understanding of the importance of the consent process | after obtaining consent for endoscopy but prior to endoscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Neilan, MT (ASCP), Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] Rozovsky FA, Consent to Treatment: A practical Guide, 4th ed. Aspen Publishers 2007
- [Background] Communicating with patients who have limited literacy skills. Report of the National Work Group on Literacy and Health. J Fam Pract. 1998 Feb;46(2):168-76. PMID 9487325
- [Result] Dewalt DA, Berkman ND, Sheridan S, Lohr KN, Pignone MP. Literacy and health outcomes: a systematic review of the literature. J Gen Intern Med. 2004 Dec;19(12):1228-39. doi: 10.1111/j.1525-1497.2004.40153.x. PMID 15610334
- [Result] Sudore RL, Landefeld CS, Williams BA, Barnes DE, Lindquist K, Schillinger D. Use of a modified informed consent process among vulnerable patients: a descriptive study. J Gen Intern Med. 2006 Aug;21(8):867-73. doi: 10.1111/j.1525-1497.2006.00535.x. PMID 16881949
- [Result] Cassileth BR, Zupkis RV, Sutton-Smith K, March V. Informed consent -- why are its goals imperfectly realized? N Engl J Med. 1980 Apr 17;302(16):896-900. doi: 10.1056/NEJM198004173021605. PMID 7360175
- [Result] Lavelle-Jones C, Byrne DJ, Rice P, Cuschieri A. Factors affecting quality of informed consent. BMJ. 1993 Apr 3;306(6882):885-90. doi: 10.1136/bmj.306.6882.885. PMID 8490411